CLINICAL TRIAL: NCT07111650
Title: Relationship Between Pelvic Floor Muscle Activity and Voice Acoustic Parameters in Young Adults
Brief Title: Relation of Pelvic Floor Muscle and Phonation
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Sponsor
Other Study IDs: PFM_PHONATION
Record Dates: First submitted 2025-04-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: acoustic analysis; Electromyography; Pelvic floor muscle; phonation; Voice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trunk is divided into the thoracic cavity above and the abdominal cavity below by the thoracic diaphragm. The vocal cords are located in the upper region of the thoracic cavity, in the area between the folds known as the larynx. The pelvic floor is a multilayered muscular sling that is located in the lower part of the abdomen. There is a relationship between the pelvic floor and the larynx through fascial connections along the trunk .

Pelvic floor muscles (PFM) play an important role in bowel and bladder continence, sexual function, lift abdominal and pelvic organs, regulation of intra-abdominal pressure and maintenance of respiration and posture. The larynx has many important functions such as protecting the airway, facilitating natural breathing, producing phonation or sound, increasing intra-abdominal pressure during straining, defecation, micturition and labour. Structural integrity and functionality between the respiratory, laryngeal or phonation levels and the resonant cavities are essential for correct voice production. The pelvic floor, thoracic diaphragm and larynx move simultaneously caudally when inhaling and cranially when exhaling, like a piston.

Voice is produced by the larynx during expiration when air passes through the trachea, setting the vocal cords into vibration. The tension of the vocal cords and sufficient subglottal pressure are essential for phonation. Additionally, the abdominal muscles play a crucial role in controlling the expiratory phase of speech by counteracting the recoil pressures of the lungs. This allows for the production of longer utterances and the maintenance of subglottal pressure throughout phonation.Voice hygiene and proper breathing techniques are crucial for both professional and non-professional voice users such as singers, academics, call center employees, and religious leaders. Healthy sound production requires PFM stability, balanced abdominal muscles, and effective respiratory control

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer
* Age between 18- 40 years

Exclusion Criteria:

1. urological, gynecological, respiratory, or vocal disorders,
2. cognitive or perceptual problems,
3. being pregnant,
4. being in the premenstrual or menstrual phase on the evaluation day,
5. having allergies, cold, or flu on the evaluation day,
6. perineal sensitivity,
7. any surgery in the abdominal, stomach, respiratory, laryngeal, and/or head and neck regions,
8. vocal complaints for at least 15 days,
9. hearing complaints.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle activity | Baseline
  Pelvic floor muscle strength and endurance were assessed using the Neurotrac® Myoplus 2 Pro two-channel EMG Biofeedback device. One channel's electrodes were placed in the anal region to assess the pelvic floor muscles, while the other channel's electrodes were placed on the transversus abdominis, with a reference electrode located on the thigh. Initially, the participant was instructed on how to contract and relax the pelvic floor muscles, followed by a trial period.
Acoustic Voice Analysis | Baseline
  Both the recordings and the analyses were performed in the same laboratory using the Kay Elemetrics Computerised Speech Lab (CSL) KayPENTAX Model 4500 system. Recordings were made using a KayPENTAX CSL Model 4500 unit and a Shure SM48 microphone connected to a desktop computer. Participants were seated on a chair in front of the computer, and the microphone was positioned at a 45-degree angle, 10 cm away from the speaker's mouth. All recordings were saved in the CSL programme as sound files (nsp) with a sampling rate of 44.01 kHz and a resolution of 24-bits. Data analyses were performed on the same computer and device. Participants were instructed to produce a natural and relaxed /a/ phonation without straining or raising their voice, similar to how they normally speak in daily life.

SECONDARY OUTCOMES:
Maximum phonation time | Baseline
  Voice recordings for maximum phonation time (MPT) were recorded using the CSL device, and analyses were performed on the same system. For the MPT, participants were instructed to take a deep breath and produce a long /a/ phonation at a normal pitch and loudness until they ran out of breath, without holding or pausing their breath. This measurement was repeated three times, and the average duration across the three trials was calculated in seconds.
s/z ratio | Baseline
  Voice recordings for the s/z ratio were recorded using the CSL device, and analyses were performed. For the s/z ratio, participants were asked to take a deep breath and produce a long /s/ phonation at a normal pitch and loudness until they ran out of breath. The entire procedure was repeated three times. They were instructed to perform the same process three times with the /z/ phonation. After calculating the maximum duration of both /s/ and /z/ phonations, the s/z ratio was determined by dividing the maximum /s/ duration by the maximum /z/ duration.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kutahya Health Sciences University, Kütahya, Merkez
  - Kutahya Helath Sciences University- Health Sciences Faculty, Kütahya, Merkez

IPD SHARING:
Plan to Share IPD: Undecided